CLINICAL TRIAL: NCT05159414
Title: A Single Center, Open-label, Exploratory Study to Evaluate the Efficacy and Safety of the Application of Pulse Electrical Stimulation Around the Eye in Glaucoma Patients
Brief Title: Study of Application of Pulse Electrical Stimulation Around Eye in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NE_RTN_001
Record Dates: First submitted 2021-11-02; First posted 2021-12-16 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glaucoma patients (Experimental): Duration of study period(per participant): Screening period(0-4weeks), Intervention period(16weeks) Patient needs to visit site at least 5 times(Screening, V2, V3, V4, V5). V2 can be done with screening visit. Visit 3, 4, 5 is 2weeks, 6weeks, and 16weeks after visit 2(Baseline).
  Interventions: Device: Pulse Electrical Stimulation

INTERVENTIONS:
Device: Pulse Electrical Stimulation — Pulse Electrical Stimulation Patients wear our clinical trial device 30mins once a day for 16weeks.

SUMMARY:
This study aims to evaluate the efficacy and safety of applying pulse electrical stimulation around eyes of glaucoma patients.

DETAILED DESCRIPTION:
Duration of study period(per participant): Screening period(0-4weeks), Intervention period(16weeks) Patient needs to visit site at least 5 times(Screening, V2, V3, V4, V5). V2 can be done with screening visit. Visit 3, 4, 5 is 2weeks, 6weeks, and 16weeks after visit 2(Baseline).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 19 to 75 years of age, at the time of screening
* Patients with normal tension glaucoma or open angle glaucoma
* Patients with best-corrected visual acuity of 20/40 or more
* Patients whose Mean Deviation(MD) value of visual field test is -6dB or less
* Patients who have stable eye pressure of less than 20mmHg over the past 2 months
* If glaucoma treatment is in progress, the type, dose, and form of drug for treatment are stable for more than 2 months
* A person who has no pregnancy plan during the clinical trial period and has agreed to an effective contraceptive plan for WOCBP(Women of child bearing potential)

  * WONCBP(Women of non-child bearing potential) must meet at least one of the following criteria:

    1. Postmenopausal women who are at least 45 years old and had no menses for 24 consecutive months
    2. A woman who underwent hysterectomy of bilateral ovarian resection recorded by a doctor
  * All other female patients will be considered WOCBP.
* A person who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

* Ophthalmological and neurological diseases that can affect visual field test(e.g., optic neuritis, diabetic retinopathy, age-related macular degeneration, and the epiretinal membrane)
* A person with a history of surgery related to eyeball excluding simple cataract surgery or orbital surgery such as orbital fracture
* Those who have more than -6D of refractive errors
* Those who have cataracts of ETDRS(Early Treatment Diabetic Retinopathy Study) grade 3 or higher
* Those who have a history of trauma around the eyeball, such as an orbital fracture, etc.,
* Patients with active malignancy or history of malignancy, except completely treated in situ carcinoma of the cervix, completely treated and resected non-metastatic squamous of basal cell carcinoma of the skin.
* A person who recently(within 1 month before the clinical trial medical device is applied) suffered severe trauma or underwent major surgery
* Pregnant or lactating women
* Any other severe acute or chronic medical or psychological conditions
* Those who can't understand or read the consent form of this clinical trial(e.g. illiterate or foreigners)
* Any other cases that PI considers hard to participate in this clinical trial(e.g. heart-related problems, seizure, epilepsy. Patients transplanted metal or electronic device in head & neck. Patient suffering from unknown pain. Patients who are warned not to use out clinical trial device or is prohibited from using it.)
* In the case of participating in other clinical trials within 6 months prior to the time of obtaining the consent form
* Subjects who are not suitable for the clinical trial, are likely to be in danger when participate in the study or interfere with the interpretation of the trial results.
* Brain and neck implant or pacemaker including deep brain stimulation device. Implantable or wearable cardioverter defibrillator. (Dental implants are accepted.)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure | baseline, 2, 6, 12, 16 weeks
  Check the change of intraocular pressure in the baseline, 2, 6, 12, 16 weeks
Changes in visual acuity | baseline, 2, 6, 12, 16 weeks
  Check the change of visual acuity in the baseline, 2, 6, 12, 16 weeks
Changes in mean deviation (MD) | baseline, 2, 6, 12, 16 weeks
  Check the change of mean deviation(MD) in the baseline, 2, 6, 12, 16 weeks
Changes in pattern standard deviation(PSD) | baseline, 2, 6, 12, 16 weeks
  Check the change of pattern standard deviation(PSD) in the baseline, 2, 6, 12, 16 weeks
Changes in visual field index(VFI) | baseline, 2, 6, 12, 16 weeks
  Check the change of visual field index(VFI) in the baseline, 2, 6, 12, 16 weeks

SECONDARY OUTCOMES:
Changes in parapapillary retinal nerve fiber layer thickness (RNFLT) using optical coherence tomography(OCT) | baseline, 6, 16 weeks
  Check the change of parapapillary retinal nerve fiber layer thickness(RNFLT) in the baseline, 6, 16 weeks
Changes in Laminar cribrosa (LC) depth using optical coherence tomography(OCT) | baseline, 6, 16 weeks
  Check the change of Laminar cribrosa(LC) depth in the baseline, 6, 16 weeks
Changes in macular ganglion cell-inner plexiform layer thickness (GCIPLT) using optical coherence tomography(OCT) | baseline, 6, 16 weeks
  Check the change of macular ganglion cell-inner plexiform layer thickness(GCIPLT) in the baseline, 6, 16 weeks
Changes in circumpapillary vessel density (cpVD) using Optical coherence tomography angiography(OCT-A) | baseline, 6, 16 weeks
  Check the change of circumpapillary vessel density(cpVD) in the baseline, 6, 16 weeks
Changes in macular vessel density (mVD) using Optical coherence tomography angiography(OCT-A) | baseline, 6, 16 weeks
  Check the change of macular vessel density(mVD) in the baseline, 6, 16 weeks
Changes in N95 amplitude using pattern Electroretinogram(ERG) | baseline, 6, 16 weeks
  Check the change of N95 amplitude in the baseline, 6, 16 weeks
Changes in N95 latency using pattern Electroretinogram(ERG) | baseline, 6, 16 weeks
  Check the change of latency in the baseline, 6, 16 weeks
Changes in Glaucoma Quality of Life-15 (GQL-15) | baseline, 6, 16 weeks
  Check the change of Glaucoma Quality of Life-15(GQL-15) score in the baseline, 6, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Youn Hye Jo, Ph. D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Department of Ophthalmology, Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No